CLINICAL TRIAL: NCT03299387
Title: INtravesical Antimicrobial Agents Versus STANDard Oral Antibiotics for the Treatment of Acute Urinary Tract Infection in Women With Recurrent Urinary Tract Infection (INSTANT Study)
Brief Title: INtravesical Antimicrobial Agents v STANDard Oral Antibiotics for the Treatment of Acute UTI in Women With rUTI
Acronym: INSTANT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never recruited
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deborah J. Lightner, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-002887
Record Dates: First submitted 2017-09-20; First posted 2017-10-03 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Urinary Tract Infections
Keywords: urinary tract; infection; recurrent; women
MeSH Terms: conditions — Urinary Tract Infections; Infections; Recurrence | interventions — Nitrofurantoin; Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Nitrofurantoin (Active Comparator): Participants will randomized to oral nitrofurantoin
  Interventions: Drug: Nitrofurantoin
- Intravesical Gentamicin (Active Comparator): Participants will be randomized to intravesical gentamicin
  Interventions: Drug: Gentamicin

INTERVENTIONS:
Drug: Nitrofurantoin — Participants will receive oral Nitrofurantoin 100 mg twice daily for 7 days
  Other Names: Macrobid, Furadantin, Macrodantin
  Arms: Oral Nitrofurantoin
Drug: Gentamicin — Participants will receive intravesical via catheter Gentamicin solution 25 mg in 50cc for 3 days
  Other Names: Gentak, Garamycin
  Arms: Intravesical Gentamicin

SUMMARY:
Women have problems with oral antibiotics, including vagina and bowel infections. Also, bacteria causing urinary infections are becoming more resistant to oral antibiotis. Placement of antibiotic directly into the bladder does not cause these problems and are at doses that are may be able to stop bacteria from being resistant to antibiotics.

DETAILED DESCRIPTION:
Each participant once enrolled returns with an active Urinary Tract Infection (UTI), confirmed by urine void. Participants will complete an UTI questionnaire, and if consistent with a simple non-febrile UTI will be randomized to one of two arms: oral nitrofurantoin treatment for 7 days, or intravesical gentamicin instillation once a day for three days. Patients will be followed for symptom relief with a repeat voided urine in 7 to 10 days, and with a repeated questionnaire for symptom relief.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand study procedures and to comply with them for the entire length of the study.

Exclusion Criteria:

* Patients who report that they are pregnant.
* Patients with a positive urine pregnancy test
* Patients with a history of renal transplantation.
* Patients with bladder augmentation procedures using bowel.
* Patients with poorly controlled Type II diabetes, Hgb A1C >6.5%
* Patients with spinal cord injury, ASIA Impairment Scale of C or higher.
* Patients with pelvic surgery within 6 months.
* Patients with urologic procedure within 6 months.
* Patients with a history of reconstructive urologic surgery, such as reflux, congenital abnormality.
* Immunocompromised patients being treated for malignancy or a history of actively treated malignancy within 5 years.
* Patients with active systemic autoimmune disease.
* Patients on systemic immunosuppression.
* Use of antibiotic prophylaxis within 6 months
* Use of antibiotics within 10 days of active infection
* Allergy/sensitivity to gentamicin or nitrofurantoin.
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual to give written informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Premenopausal or perimenopausal healthy female patients with an active urinary tract infection and at least two symptomatic and culture-proven urinary tract infections within the past 12 months
Enrollment: 0 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Change in microbiologic effect of a chronic acute Urinary Tract Infection | baseline, 7-10 days
  Microbiological culture growth of susceptible organisms obtained on day 0, compared with voided urine culture as no growth in 24-48 hours obtained at 7-10 days
Change in symptomatic relief of a chronic acute Urinary Tract Infection | baseline, 7-10 days
  Completion of a Symptom Urinary Tract Questionnaire. Tracking the symptoms in the past 24 hours. Indicating how severe and how bothersome they were. Severe ranging from 0 (Did not have) to 3 (Severe). Bothersome ranging from 0 (Not at all) to 3 (A lot)

SECONDARY OUTCOMES:
To establish the clinical FTE needs for providing urgent intravesical treatments | baseline, through stufy completion, an average of one year
  Nursing needs to provide intravesical treatments of acute Urinary Tract Infections (UTI) in women with chronic recurrent UTIs. Measured in amount of participants and FTE requirement for nursing staff.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Lightner, MD, Principal Investigator — Mayo Clinic; Audrey N Schuetz, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials